CLINICAL TRIAL: NCT00894530
Title: The Effects of Azithromycin Ophthalmic Solution, 1% Versus Placebo in Subjects With Blepharitis During a Four-Week Treatment Period (P08638)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P08638; 044-102
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-10

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Azithromycin ophthalmic solution, 1%
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin ophthalmic solution, 1% — One drop in each eye twice a day for the first two days; then one drop in each eye once a day for 26 days
  Arms: 1
Drug: Placebo — One drop in each eye twice a day for the first two days; then one drop in each eye once a day for 26 days
  Arms: 2

SUMMARY:
The objective of this study is to compare the safety and efficacy of azithromycin ophthalmic solution, 1% versus placebo over a four-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have best corrected visual acuity in both eyes of at least +0.7 or better
* If female, are non-pregnant or non-lactating
* Have a current diagnosis of blepharitis in one or both eyes

Exclusion Criteria:

* Have lid structural abnormalities
* Have suspected ocular fungal or viral infection
* Have practiced warm compress therapy within 14 days prior to Visit 2
* Unable to withhold the use of contact lenses during the treatment or follow-up periods
* Unable to withhold the use of ocular cosmetic products within 24 hours prior to study visits
* Have had penetrating intraocular surgery within 90 days prior to Visit 2
* Have had ocular surface surgery within the past year prior to Visit 2
* Have a serious medical condition which could confound study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Eyelid margin erythema | Four weeks

SECONDARY OUTCOMES:
Signs and symptoms of Blepharitis | One week, two weeks, three weeks, four weeks, six weeks, eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD,PhD, Study Chair — Medical Monitor, Inspire
Locations (26):
- United States (26):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - McDonald Eye Associates, Fayetteville, Arkansas
  - Sall Research Medical Center, Inc., Artesia, California
  - Sall Research Medical Center, Artesia, California
  - United Medical Research Company, Inglewood, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Coastal Vision Medical Group, Newport Beach, California
  - West Coast Eye Care, San Diego, California
  - Hernando Eye Institute, Brooksville, Florida
  - Center for Excellence in Eye Care, Miami, Florida
  - Wohl Eye Center, Bloomingdale, Illinois
  - Thomas John Vision Institute, Tinley Park, Illinois
  - Grene Vision Group, Wichita, Kansas
  - Taustine Eye Center, Louisville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care Ltd, Washington, Missouri
  - David M. Ringel, DO, PA, Sewell, New Jersey
  - Brar-Parekh Eye Associates, Woodland Park, New Jersey
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Park Ophthalmology, Durham, North Carolina
  - Ohio State University - College of Optometry, Columbus, Ohio
  - Columbus Ophthalmology Associates, Columbus, Ohio
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - Total Eye Care, PA, Memphis, Tennessee
  - Eye Clinics of South Texas, San Antonio, Texas